CLINICAL TRIAL: NCT00809081
Title: A Prospective, Randomized Trial of Early Enteral Feeding After Pylorus Preserving Pancreatoduodenectomy
Brief Title: Early Enteral Feeding After Pylorus Preserving Pancreatoduodenectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Dong Sup Yoon/Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN Vs PN
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Pancreas Cancer; Bile Duct Cancer; Ampulla of Vater Cancer
Keywords: periampullar carcinoma; Pancreaticoduodenectomy; Enteral feeding; Total Parenteral Support
MeSH Terms: conditions — Pancreatic Neoplasms; Bile Duct Neoplasms | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): 1. Enteral Feeding
  Interventions: Procedure: Enteral Feeding and Total Parental Support
- 2 (No Intervention): Total Parental support
  Interventions: Procedure: Enteral Feeding and Total Parental Support

INTERVENTIONS:
Procedure: Enteral Feeding and Total Parental Support — Enteral Feeding : 20ml/hr on POD1
  * Velocity is progressively increased by 20ml/d until full nutritional goal (25Kcal/Kg)
  Other Names: Total Parental support: 1000 kcal /d on POD 1; : Velocity is progressively increased by 20ml/d; until full nutritional goal (25Kcal/Kg)

SUMMARY:
Pancreaticoduodenectomy is associated with a high incidence of postoperative complications. These postoperative complications could delay postoperative resumption of adequate oral intake. Clinical study on postoperative feeding after pancreaticoduodenectomy is very limited. Method of Nutritional support (Enteral feeding or total parenteral support)after pancreaticoduodenectomy is controversial.

1. To evaluate whether early enteral nutrition may be a suitable alternative to total parenteral nutrition
2. To evaluate whether enteral feeding improve nutritional status after pancreaticoduodenectomy

DETAILED DESCRIPTION:
Pancreaticoduodenectomy is associated with a high incidence of postoperative complications. These postoperative complications could delay postoperative resumption of adequate oral intake. The use of TPN significantly increases postoperative complications, especially those associate with infections. However, method of Nutritional support (Enteral feeding or total parenteral support)after pancreaticoduodenectomy is controversial.

1. To evaluate whether early enteral nutrition may be decreased the postoperative complications
2. To evaluate whether enteral feeding improve nutritional status after pancreaticoduodenectomy
3. To determine the optimal method for postoperative nutritional support

ELIGIBILITY:
Inclusion Criteria:

* Periampullar carcinoma
* Pancreaticoduonectomy
* KARNOFSKY PERFORMANCE SCALE > 70
* No history of Major operation

Exclusion Criteria:

* Creatinine level>3mg/L
* Ascitis/portal hypertension
* New York Heart Association class>3
* COPD
* Preoperative Radiotheraly/chemotherapy
* Unresectable primary cancer
* Palliative surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-06 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of early postoperative enteral feeding | Postoperative 21 days

SECONDARY OUTCOMES:
To evaluate the nutritional status | Postoperative 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sup Yoon, MD,PhD, Principal Investigator — Yonsei University
Locations (1):
- Yongdong Severance Hospital, Seoul, South Korea